CLINICAL TRIAL: NCT03890263
Title: Evaluating the Outcomes and Experiences of Chronic Pain Self-Management Support with an Opioid De-prescribing Intervention: a Mixed Methods Study
Brief Title: Evaluating Chronic Pain Self-Management Support with an Opioid De-prescribing Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jordan Miller, PT, PhD, Assistant Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 373022
Record Dates: First submitted 2019-03-21; First posted 2019-03-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This study will use parallel mixed methods including:
  1. An interrupted time series design to evaluate outcomes of an evidence-based self-management intervention and opioid deprescribing. This time series will include 18 assessments over 36-weeks from 12 weeks prior to implementation of the combined intervention to 24 weeks after implementation of the combined intervention.
  2. Qualitative semi-structured interviews informed by an interpretive description approach with patients and health care providers to understand their perspectives and experiences.
  3. A nested cross sectional evaluation to determine the characteristics of people who are identified on high doses of opioids in primary care in South Eastern Ontario. Characteristics collected will include: age, sex, gender, education, household income, postal code/geographic location, work status, caregiver status, early childhood trauma, depression, post-traumatic stress, health-related quality of life, and comorbidities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Opioid deprescribing and self-management (Experimental)
  Interventions: Behavioral: Chronic Pain Self-Management Support

INTERVENTIONS:
Behavioral: Chronic Pain Self-Management Support — Family physicians and nurse practitioners will participate in an academic detailing session with a pharmacist that focuses on safe, evidence-based opioid deprescribing. The pharmacist will provide pre-visit recommendations for each visit with a person on high doses of opioids. The pharmacist and healthcare providers will develop a patient centered, opioid taper schedule, with follow-up at 2 to 4 week intervals to assess for efficacy and safety.
  The self-management intervention will be "Chronic Pain Self-management Support with Pain Science Education and Exercise" (COMMENCE), which consists of 2 visits per week over 6 weeks. One visit per week is 1.5 hours in a group format. with education about self-management and pain science as well as cognitive behavioural principles. The 2nd visit each week is 30 minutes in a one-to-one format and is individually tailored to support implementation of self-management plans and development of an exercise program.
  Other Names: Opioid De-prescription

SUMMARY:
This study will evaluate the outcomes of the combination of chronic pain self-management support with opioid deprescription, improve our understanding of the experiences and perspectives of patients and healthcare providers with this approach, and determine the characteristics of people on opioids in primary care to inform future research and implementation of this approach

DETAILED DESCRIPTION:
Chronic pain is a burden on individuals, the health system, and society. Opioid prescriptions have increased over three decades with the aim of reducing the burden of chronic pain. Unfortunately, increases in opioids have not improved functional outcomes for people with pain and opioid related side-effects and deaths have accompanied the rise in use. Opioid deprescribing (reducing the dose or transitioning off of opioids) has the potential to improve health outcomes for people on opioids for chronic pain. One of the evidence based approaches to deprescribing includes providing an interdisciplinary pain program for individuals to help manage their pain as they reduce their dose or transition off of opioids.

Unfortunately, the inability to access multidisciplinary pain programs is a barrier faced by most people living with pain and their primary care providers. Self-management support has been shown to improve pain and function for people with chronic pain and may be more feasible to offer in primary care to support people as they try to reduce their dose or transition off of opioids. Evidence on the outcomes of pairing self-management support with opioid deprescribing is lacking, however. This study will evaluate the outcomes of the combination of chronic pain self-management support with opioid deprescription, improve our understanding of the experiences and perspectives of patients and healthcare providers with this approach, and determine the characteristics of people on opioids in primary care to inform future research and implementation of this approach. If effective, this approach could be implemented more widely. The results of this study, therefore, have the potential to improve health outcomes for people taking opioid medications for chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain for >3months
* On opioid medications with a dose of at least 50 milligram morphine equivalents per day
* Ability to communicate effectively using the English language, including reading and writing

Exclusion Criteria:

- Chronic pain due to cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Changes in Opioid Use | Every 2 weeks for 36 weeks
  Changes in opioid use will be measured using milligram morphine equivalents per day. This will be collected every two weeks throughout the 36-week study period.
Changes in Pain Severity: Pain Severity Scale of the Brief Pain Inventory (BPI) | Every 2 weeks for 36 weeks
  Changes in pain severity will be measured using the Pain Severity Scale of the Brief Pain Inventory (BPI), which asks about the participant's pain at its worst, at its best, on overage and right now. It uses an 11-point scale ranging from 0 to 10, where 0 indicates no pain at all and 10 indicates the worst pain imaginable. The mean severity of all four individual scores will be used for the main analysis (total of all four scores divided by four). Pain severity will be assessed every two weeks, measuring the change across the course of the study.
Changes in Pain Interference: Pain Interference Scale of the Brief Pain Inventory (BPI) | Every 2 weeks for 36 weeks
  Changes in pain interference will be measured with the Pain Interference Scale of the Brief Pain Inventory (BPI), which uses an 11-point scale to measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. On the scale, 0 indicates that pain has not interfered with the activity at all and 10 indicates that pain has completely interfered with the activity. BPI Pain Interference will scored as the mean of the scores on seven interference items (total of all seven scores divided by seven). Pain interference will be assessed every two weeks, measuring the change across the course of the study.
Occurrence of Adverse Events | Every 2 weeks for 36 weeks
  Occurrence adverse events over a 36 week period will be recorded using an adverse events questionnaire that is consistent with reporting guidelines and asks: 1) if the patient has experienced any events as a result of any of the treatments received (yes/no); 2) what adverse events were experienced (choose from a drop-down list or 'other'); 3) how long the event lasted (hours or days); 4) How severe the adverse event was (0-10 scale, where 0 indicates not severe at all and 10 indicates very severe). Each occurrence (the type of adverse event and duration and severity) will be recorded individually for reporting purposes as well as descriptive purposes.

SECONDARY OUTCOMES:
Adverse Childhood Experiences (ACE) Questionnaire | Baseline
  The Adverse Childhood Experiences (ACE) Questionnaire will be used to identify adverse childhood experiences. It has shown good reliability and predictive validity. Several studies have demonstrated its ability to predict the onset of chronic pain in adults and it has been shown to be associated with initiation of opioid use, opioid dependence, opioid misuse, and likelihood of experiencing an opioid overdose. The questionnaire has 10 questions about various stressful childhood experiences. For each question an answer of No = 0 and and answer of Yes = 1. The total score out of 10 possible points will be used. This questionnaire will be administered only once at baseline.
9-item Patient Health Questionnaire (PHQ-9) | Baseline
  The PHQ-9 demonstrates good reliability and validity and will be used to screen for depression using a cut-score of 10 points as has been suggested in the literature. The PHQ-9 has 9 questions, which all start with, "Over the past two weeks, how often have you been bothered by the following problem...:" The participant answers each one on a four-point Likert Scale, where 0 indicates not bothered at all and 3 indicates bothered nearly every day. The total score out of a possible 27 points will be used. This questionnaire will be administered only once at baseline to describe the population.
Post-traumatic Stress Disorder (PTSD) Checklist - Civilian Version | Baseline
  The PTSD Checklist - Civilian Version will be used to identify the presence and severity of post-traumatic stress symptoms. The checklist has 17 questions. The instructions begin with: "Below is a list of problems and complaints that people sometimes have in response to stressful life experiences. Please read each one carefully, then pick the answer that indicates how much you have been bothered by that problem in the last month." The answers are on a five-point scale, where 1 indicates not bothered at all and 5 indicates extremely bothered. The total severity score out of a possible 85 points will be used. A score range of 17-29 shows little to no severity; a score range of 28-29 shows some PTSD symptoms; a score range of 30-44 shows moderate to moderately high severity of PTSD symptoms; and a score range of 45-85 shows high severity of PTSD symptoms. This questionnaire will be administered only once at baseline to describe the population
Health-related Quality of Life: EuroQOL-5D (EQ-5D-5L) | Baseline
  Health-related quality of life will be measured with the EuroQOL-5D (EQ-5D-5L). This questionnaire has two parts: the first is the 5-question 'descriptive system', which asks respondents to 'select the ONE statement that BEST describes your health TODAY' for 5 health dimensions: mobility, self care, usual activities, pain/discomfort, anxiety/depression. The 5 statements for each dimension are "no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems (5)". The 5 answers form a 5-digit code describing the respondent's 'health state'. Eg. the health state '12345' indicates no problems with mobility, slight problems with washing/dressing, moderate problems with usual activities, severe pain or discomfort and extreme anxiety or depression.
  The second part asks respondents to rate their global health today on a visual analogue scale from 0-100, where 100 means the best health imaginable and 0 means the worst health imaginable.
Change in patient specific functional scale (PSFS) | Baseline, 12 weeks, 36 weeks
  Changes in function will be measured with the Patient-Specific Functional Scale. Participants are asked to identify three important activities that they are having difficulty doing or are unable to do as a result of their primary condition. For each activity, they are asked to use an 11-point scale to rate their difficulty, where 0 indicates they are able to perform activity at the same level as before the injury or problem (No issues) and 10 indicates they are unable to perform activity (Cannot perform). The mean score will be used (sum of the activity scores divided by the number of activities). Minimum detectable change (90%CI) for average score = 2 points. The same activities will be rated at baseline, 12 weeks and 36 weeks, and the changes in mean scores between time points will be recorded.
Global Rating of Change in function (12-weeks) | 12-weeks
  Changes in Global Rating of Change in Functional Abilities will be measured using an 11-point scale ranging from -5 (much worse) to +5 (completely recovered) as has been recommended in the literature for self-reported rating of change. This will be measured at 12 weeks and 36 weeks, recording the change across time points.
Global Rating of Change in function (36-weeks) | 36 weeks
  Changes in Global Rating of Change in Functional Abilities will be measured using an 11-point scale ranging from -5 (much worse) to +5 (completely recovered) as has been recommended in the literature for self-reported rating of change. This will be measured at 12 weeks and 36 weeks, recording the change across time points.
Goal Attainment Scale (12-weeks) | 12-weeks
  Changes in the attainment of three stated functional goals will be measured using the Goal Attainment Scale. This is a 5-point scale, used to assess attainment of individual goals, ranging from -2 to +2, where -2 indicates a level of attainment much less than expected, 0 indicates the expected level of attainment, and +2 indicates a level of attainment much more than expected. The mean score will be used (sum of the attainment scores divided by the number of attainment scores). The goals will be identified at baseline and goal attainment will be measured at 12 weeks and 36 weeks.
Goal Attainment Scale (36-weeks) | 12-weeks and 36 weeks
  Changes in the attainment of three stated functional goals will be measured using the Goal Attainment Scale. This is a 5-point scale, used to assess attainment of individual goals, ranging from -2 to +2, where -2 indicates a level of attainment much less than expected, 0 indicates the expected level of attainment, and +2 indicates a level of attainment much more than expected. The mean score will be used (sum of the attainment scores divided by the number of attainment scores). The goals will be identified at baseline and goal attainment will be measured at 12 weeks and 36 weeks.
Satisfaction with care (12-weeks): 11-point scale | 12-weeks
  Satisfaction with Care will be measured using an 11-point scale ranging from -5 (very dissatisfied) to +5 (very satisfied) as has been recommended in the literature for self-reported rating of change. This will be measured this at 12 weeks and 36 weeks.
Satisfaction with care (36-weeks): 11-point scale | 36-weeks
  Satisfaction with Care will be measured using an 11-point scale ranging from -5 (very dissatisfied) to +5 (very satisfied) as has been recommended in the literature for self-reported rating of change. We will measure this at 12 weeks and 36 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Queen's University
Locations (1):
- Queen's Family Health Team, Belleville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No